CLINICAL TRIAL: NCT03016039
Title: Curcumin Supplementation for Gynecological Diseases Including Pelvic Inflammatory Disease Endometritis, Endometriosis: A Pilot Study
Brief Title: Curcumin Supplementation for Gynecological Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0210-16-MMC
Record Dates: First submitted 2016-12-11; First posted 2017-01-10 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Curcumin Use for Gynecological Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary supplementation (Experimental): This group will receive Dietary supplementation
  Interventions: Dietary Supplement: Curcumin supplementation
- conventional treatment (No Intervention): conventional Antibiotic treatment without curcumin supplementation

INTERVENTIONS:
Dietary Supplement: Curcumin supplementation — use of curcumin supplementation as an additive treatment to the conventional treatment
  Arms: Dietary supplementation

SUMMARY:
To use curcumin supplementation as an additive treatment to induce clinical, biochemical response and remission in patients with suspected Pelvic inflammatory disease, Tubo ovarian abcess, Endometritis, wound infection.

Hypothesis: An addition of oral curcumin to highly suspected PID/Endometritis/Wound infection patients may augment clinical and biochemical response and accelerates the improvements of the sign symptoms and reported outcomes of those diseases.

DETAILED DESCRIPTION:
Pelvic inflammatory disease (PID), Endometritis, Wound infection are infections of the female reproductive system. Although PID is a well known pathophysiology the diagnosis method I not well established and its true magnitude is unknown. Many women report that they have been treated for PID when they did not suffer from it and vice versa. Hence the main way to diagnose remains clinical and currently there is no well-established biochemical marker. In endometritis and wound infection the cause may be known but the pathogens involved in the disease formation vary as for this broad spectrum antibiotic is needed.

Aims: To use curcumin supplementation as an additive treatment to induce clinical, biochemical response and remission in patients with suspected PID, Tubo ovarian abcess, Endometritis, wound infection.

Hypothesis: An addition of oral curcumin to highly suspected PID/Endometritis/Wound infection patients may augment clinical and biochemical response and accelerates the improvements of the sign symptoms and reported outcomes of those diseases.

Rational: Curcumin treatment has been shown to safe and efficient in inflammatory states such as in mild-moderate Ulcerative colitis (UC), obesity, and type II diabetes mellitus when used as an add-on to conventional treatment.

In the gynecology and especially in the PID/Tubo ovarian abcess diseases the use of Curcumin as a supplement has never been studied.

In the future it is necessary to study the use of curcumin in different gynecological diseases (e.g Endometriosis/Premenstrual syndrome (PMS) and also in gynecology oncology) in which inflammatory and immune response are involve in the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* The patient was admitted with a diagnosis of Pelvic inflammatory disease / Tubo ovarian abcess, surgical wound infection, Endometritis
* No Antibiotic treatment was given prior to her recruitment for the study
* The women is not in menopause

Exclusion Criteria:

* Age below 18 and above 52
* Antibiotic treatment was given prior to her recruitment for the study
* The women is in menopause
* Pregnant women. Known other inflammatory disease.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-01-07; Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Change in the Levels of C reactive protein | at recruitment and after two week and after one month
Change in the Levels of White blood cells | at recruitment and after two week and after one month

CONTACTS AND LOCATIONS:
Locations (1):
- Meir hospital, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No